CLINICAL TRIAL: NCT05158920
Title: Randomized Controlled Trial Investigating the Effectiveness of Mindfulness-Based Cognitive Therapy for Suicidal Patients
Brief Title: A Mindfulness-Based Cognitive Therapy for Suicidal Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC/20160609/MBCT
Record Dates: First submitted 2021-12-02; First posted 2021-12-15 (Actual); Last update posted 2022-01-10 (Actual); Status verified 2021-12

CONDITIONS: Suicidal Ideation; Suicide Attempt
MeSH Terms: conditions — Suicidal Ideation; Suicide, Attempted | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial comparing an experimental condition (Treatment As Usual + Mindfulness-Based Cognitive Therapy) and a control condition (Treatment As Usual)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Participants in the intervention group received Mindfulness-Based Cognitive Therapy in addition to their treatment as usual.
  Interventions: Behavioral: Mindfulness-Based Cognitive Therapy for Suicidal individuals (MBCT-S)
- Control Group (No Intervention): Participants in the control group received their treatment as usual.

INTERVENTIONS:
Behavioral: Mindfulness-Based Cognitive Therapy for Suicidal individuals (MBCT-S) — MBCT-S is a group intervention of 8 weekly sessions of 2 hours combining techniques of mindfulness with important elements of cognitive therapy (e.g. safety plan and homework).
  Arms: Intervention Group

SUMMARY:
The main goal of this study is to evaluate the effectiveness ofMindfulness-Based Cognitive Therapy aimed at reducing suicidality in adults. This will test the effectiveness by studying the effect on suicidal ideation and related outcomes, compared to Treatment As Usual. The study is a multicentre randomized controlled trial conducted in out-patient Flemish mental healthcare facilities.

ELIGIBILITY:
Inclusion Criteria:

* Speak Dutch
* Be at least 18 years old
* Have access to internet
* Be suitable for group therapy
* Have mild to severe suicidal thoughts (BSS score of minimum 1)

Exclusion Criteria:

* Conditions expected to severely hinder group participation, comprehension of the training content or adherence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2018-03-02 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Suicidal ideation: The Beck Scale for Suicide Ideation | Baseline (2 weeks before the intervention), posttest (2 months after baseline assessment), follow-up (5 months after baseline assessment)
  A 21-item self-report questionnaire to measure (the severity of) suicidal ideation in adolescents and adults. Each item is rated on a scale from 0 to 2, resulting in a total score ranging from 0 to 38, with higher scores indicating more (severe) suicidal ideation.

SECONDARY OUTCOMES:
Depressive symptoms: The second edition of the Beck Depression Inventory | Baseline (2 weeks before the intervention), posttest (2 months after baseline assessment), follow-up (5 months after baseline assessment)
  A 21-item self-report questionnaire to measure depressive symptoms and attitudes in the past week. Each item is rated on a scale from 0 to 3, resulting in a total score ranging from 0 to 63, with higher scores indicating more depressive symptoms.
Hopelessness: The Beck Hopelessness Scale | Baseline (2 weeks before the intervention), posttest (2 months after baseline assessment), follow-up (5 months after baseline assessment)
  A 20-item self-report questionnaire to measure hopelessness in adolescents and adults. Each item is rated as 'true' (score = 1) or 'false' (score = 0) for them over the past week, resulting in a total score ranging from 0 to 20, with higher scores indicating higher levels of hopelessness.
Defeat: the Defeat Scale | Baseline (2 weeks before the intervention), posttest (2 months after baseline assessment), follow-up (5 months after baseline assessment)
  A 16-item self-report questionnaire to measure defeat on a five-point Likert scale.
Entrapment: the Entrapment Scale | Baseline (2 weeks before the intervention), posttest (2 months after baseline assessment), follow-up (5 months after baseline assessment)
  A 16-item self-report questionnaire to measure entrapment on a five-point Likert scale.
Worrying: The Penn State Worry Questionnaire - past week | Baseline (2 weeks before the intervention), posttest (2 months after baseline assessment), follow-up (5 months after baseline assessment)
  A 15-item self-report questionnaire to measure worrying in the past week. Each item is rated on a 7-point Likert scale ranging from 0 ("never") to 6 ("almost always").
Mindfulness: Five Facet Mindfulness Questionnaire | Baseline (2 weeks before the intervention), posttest (2 months after baseline assessment), follow-up (5 months after baseline assessment)
  A 24-item self-report questionnaire to measure five distinct facets of mindfulness: observing, describing, acting with awareness, nonjudging and nonreactivity. Each item is rated on a 5-point Likert scale ranging from 1 ("never"/"very rarely true") to 5 ("very often"/"always true"), resulting in a total score ranging from 1 to 120.

OTHER OUTCOMES:
Treatment evaluation | Posttest (2 months after baseline assessment)
  Rating of the general training (score ranging from 0 to 10) and 10 statements about several aspects of the format, content and effect of the group treatment. Of these statements, 5 were rated on a 3-point Likert scale, and 5 on a 5-point likert scale

CONTACTS AND LOCATIONS:
Overall Officials: Gwendolyn Portzky, Prof. Dr., Principal Investigator — University Ghent
Locations (1):
- Unit for Suicide Research, Ghent University, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No